CLINICAL TRIAL: NCT04657952
Title: Sphenopalatine Ganglion Block With Adrenaline Additive for Post-Dural Puncture Headache in Orthopedic Patients: A Randomized Controlled Study
Brief Title: Sphenopalatine Ganglion Block for Post-Dural Puncture Headache in Orthopedic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hussen Gamal Almawardy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34268/11/20
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Sphenopalatine Ganglion Block; Adrenaline; Post-Dural Puncture Headache; Orthopedic; Randomized Controlled Study
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medical Treatment (paracetamol) (Active Comparator): Patients will receive paracetamol 1 gm every 6 hours daily intravenously for a day.
  Interventions: Drug: Medical Treatment
- Sphenopalatine block (Experimental): Patients will receive sphenopalatine block
  Interventions: Procedure: Sphenopalatine Ganglion Block

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — Sphenopalatine Ganglion Block will be performed by a transnasal approach. Few drops of lidocaine 2% will be instilled into both anterior nares. Then a cotton-tipped applicator soaked in 4% lignocaine & adrenaline (1 to 200000 will be passed through both the nares and the end of the applicator tip will be positioned just superior to the middle turbinate and anterior to the pterygopalatine fossa and sphenopalatine ganglion for 5 min with the patient in the supine position.
  Arms: Sphenopalatine block
Drug: Medical Treatment — Patients will receive paracetamol 1 gm 6 hours daily intravenously for a day. If adequate pain relief will not be achieved, intravenous diclofenac 75 mg twice daily will be added.
  Arms: Standard medical Treatment (paracetamol)

SUMMARY:
The aim of this study is to assess the efficacy, onset and duration of analgesia of sphenopalatine ganglion bock (SPGB) using lidocaine 4% with adrenaline as a treatment of postoperative Post dural puncture headache (PDPH) of orthopedic patients after lower limbs surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the orthopedic department
* Complaining of criteria of severe post-dural puncture headache within 7 days following subarachnoid block used for lower limbs surgeries.
* American Society of Anesthesiologists (ASA) physical status I and II.

Exclusion Criteria:

* Patient refusal or uncooperative.
* Patients with uncontrollable hypertension.
* Patient with known coagulopathy.
* Patient with nasal septal deviation, polyp, history of nasal bleeding.
* Patient with allergy to local anesthetics
* American Society of Anesthesiologists physical status>2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of analgesia demonstrated by visual analogue scale (VAS) less than 4 (effective) in the first 48 hours | 48 hours
  Efficacy of analgesia demonstrated by visual analogue scale (VAS) less than 4 (effective) in the first 48 hours.
  VAS ranges from 0 to 10; 10 with worse outcome

SECONDARY OUTCOMES:
Onset of analgesia | 48 hours
  The onset time till VAS≥ 4
Duration of analgesia | 48 hours
  Duration with VAS< 4
Adverse events | 48 hours
  Local anesthetic toxicity, hypertension, postoperative epistaxis, cheek hematoma and hypoesthesia of the palate

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request
Supporting Information: Study Protocol, SAP
Access Criteria: 3 months after completing the study